CLINICAL TRIAL: NCT00198718
Title: Vitamin A Supplementation of Breast Feeding Mothers and Their Neonates at Delivery: Impact on Mother to Child Transmission of HIV During Lactation, HIV Infection Among Women During the Postpartum Year, and Infant Mortality.
Brief Title: Single-dose Postpartum Vitamin A Supplementation of Mothers and Neonates
Acronym: ZVITAMBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); University of Zimbabwe (Other); Harare City Health Department, Harare, Zimbabwe (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other); Rockefeller Foundation (Other); BASF (Industry); SARA and Linkages Projects, Academy for Educational Development, Washington DC. (Unknown); Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: (CIDA) (R/C Project 690/M3688)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Vitamin A Deficiency; HIV
Keywords: Vitamin A supplementation; HIV; Mother to child transmission of HIV; Breastfeeding
MeSH Terms: conditions — Vitamin A Deficiency; Breast Feeding | interventions — Vitamin A; retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Infant vitamin A Mother vitamin A (Experimental): Infant received 50,000 IU vitamin A, mother received 400,000 IU vitamin A
  Interventions: Drug: Vitamin A (retinyl palmitate)
- Infant vitamin A Mother placebo (Experimental): Infant received 50,000 IU vitamin A, mother received placebo
  Interventions: Drug: Vitamin A (retinyl palmitate)
- Infant placebo, mother vitamin A (Experimental): Infant received placebo, mother received 400,000 IU vitamin A
  Interventions: Drug: Vitamin A (retinyl palmitate)
- Infant received placebo, mother received placebo (Experimental): Infant and mother received placebo
  Interventions: Drug: Vitamin A (retinyl palmitate)

INTERVENTIONS:
Drug: Vitamin A (retinyl palmitate)

SUMMARY:
The ZVITAMBO PROJECT is testing whether giving mothers and infants a single large dose of vitamin A during the immediate post partum period will reduce:

1. Infant Mortality Can oral administration of a single 50,000 IU dose of vitamin A to newborn infants, a single 400,000 IU dose of vitamin A given to their lactating mothers, or supplementation of both the mother and infant during the immediate post partum period reduce infant mortality by at least 30%?
2. Mother to Child HIV transmission during breast feeding Can oral administration of a single large dose of vitamin A given during the immediate post partum period to HIV seropositive lactating women and/or their babies reduce HIV transmission via breast feeding by at least 30%?
3. Sexually transmitted HIV infection of post partum women Can a single 400,000 IU dose of vitamin A given during the immediate post partum period to HIV seronegative women reduce their likelihood of becoming HIV infected during the post partum year by at least 25%?
4. Infant feeding in the context of HIV: An operational research study was initiated mid-way through the trial to determine how UNAIDS Guidelines on infant feeding in the context of HIV could be effectively implemented and to measure the impact of such a program on infant feeding practices and postnatal HIV transmission.

Substudies:

Random subsamples of maternal and infant blood were evaluated for anemia and iron status to determine the effect of vitamin A on hematopoiesis and serum and breast milk retinol (mothers) and modified relative dose response test (infants) to determine the effect of vitamin A on vitamin A status.

A subsample of maternal and infant blood samples were evaluated for the presence of HLA-E, HLA-G, and TAP polymorphisms and their relation to prevalent HIV infection in mothers and risk of mother to child transmission.

DETAILED DESCRIPTION:
The Zimbabwe Vitamin A for Mothers and Babies (ZVITAMBO) project was a placebo-controlled randomized trial, which enrolled 14,110 mothers and their infants within 96 hours of delivery from one of 14 hospitals and clinics in greater Harare between November 25, 1997 and January 29, 2000. Mother-baby pairs were eligible if neither had an acutely life threatening condition, the baby was a singleton with birth weight >1500 g, and the mother planned to stay in Harare after delivery. Written informed consent was obtained from the mother. Socio-economic and demographic characteristics were collected by interview and obstetric details of the pregnancy and delivery were transcribed from hospital records. Gestational age was estimated. Infant birth weight was measured using an electronic scale. Infant length, infant head circumference, and maternal arm circumference were measured. Arm circumference was measured as an indicator of maternal nutritional status rather than Body Mass Index because it is less influenced by fluid fluctuations during the immediate post partum period. Addresses were recorded for the mother's urban and rural residences (it is common for urban Zimbabweans to travel frequently to extended family rural homesteads), her place of work, her husband's place of work, and that of relative who would always know her whereabouts.

At recruitment, study nurses collected plasma and serum from mothers and babies. Maternal plasma was stored at room temperature (~20° C) and other samples in a cool box (~ 10-15° C) before being transferred to the laboratory within 2 hr of collection.

Mother-baby pairs were randomized to one of four treatment groups: mother received 400,000 IU vitamin A (as retinyl palmitate) and baby received 50,000 IU vitamin A (Aa group); mother received 400,000 IU vitamin A and baby received placebo (Ap group); mother received placebo and baby received 50,000 IU vitamin A (Pa group); and both mother and baby received placebo (Pp group). Treatment and placebo capsules appeared identical and both contained a soy oil base with vitamin E as a preservative (50 IU per maternal capsule; 10 IU per infant capsule) (Tishcon Corporation, Westbury, NY, USA).

A separate team at Johns Hopkins University prepared the study capsule packets. Study identification numbers were randomly allocated to the treatment groups by computer in blocks of 12. The numbers were printed on adhesive labels and affixed to amber-colored zip-lock plastic bags that were packed with the assigned capsules. Capsule packets were prepared separately for each of the four treatment groups, and then merged into numeric order before shipping to Zimbabwe where series of packets were distributed to each recruitment site. As each mother-baby pair was recruited, the capsules in the next sequential bag were administered, and the associated study number assigned to the pair. Lists linking the study number to the treatment were kept in sealed envelopes and encrypted computer files that were not accessible to the Zimbabwe-based study team.

Pairs were followed at 6 wk, 3 mo, and then 3 monthly up to 24 months at one of three study clinics. Home visits were attempted for defaulting pairs to either their urban or rural home anywhere within the Zimbabwe borders. We initially planned to follow all HIV-positive mothers and their infants and a ~50% random sample of HIV-negative mothers and their infants for 24 months. However, in June 2000, economic conditions necessitated discontinuing the second year of follow up. This meant that 24%, 48% and 100% of the pairs were reassigned to 24 months, >18 month, and >12 month follow up, respectively. Follow up visits included assessment of recent illness, sick clinic visits, and hospitalizations by the mother or infant; anthropometric measures, infant dietary history, maternal sexual and reproductive health practices, and blood and breast milk sampling. Free clinical care included treatment of acute infections with appropriate antimicrobial drugs, referral to government treatment facilities for suspect tuberculosis, counseling and antibiotic treatment for mastitis, and oral rehydration solution education for diarrhea. HIV-related and psychosocial counseling was available throughout the study.

For mothers and infants who died, cause of death was determined from medical records for infants who died in a hospital or from review of verbal autopsy information by a study pediatrician (infants) or study obstetrician (mothers), who were masked to treatment group, for infants dying at home. Multiple causes of death were permitted and were not ranked hierarchically, in keeping with the recommendations of an expert group convened by the World Health Organization.

Maternal plasma were tested for HIV at baseline by two ELISA tests run in parallel, and by Western Blot when duplicate pairs of ELISA test results were discordant. Mothers who tested negative at baseline were retested for HIV at every blood sampling. Quality control was monitored by use of kits controls, inclusion of an internal QC sample on every plate, and participation in the quality assurance program for HIV testing of the Zimbabwe Ministry of Health. Serum retinol concentration was measured in a subsample of mothers and babies by HPLC; quality control was monitored by inclusion of standards provided by the National Institute of Standards and Technology (Gaithersburg, MD, USA) and participation in their quality assurance program Hemoglobin was measured for women enrolled from October 1, 1998 to the end of the study (about 60% of the total sample) by HemoCue (Mission Viejo, CA). Among mothers who were HIV-positive at recruitment, CD4 cells were enumerated within 48 hours of phlebotomy (Facscount, Becton Dickinson International, Erembodegem, Belgium), and viral load was measured in a subsample (Roche Amplicor HIV-1 Monitor test version 1.5, Roche Diagnostics, Alameda, CA, USA).

Plasma and cell pellets were archived from HIV-exposed infants at all visits. After follow-up was completed, the last available specimen from each infant was tested (plasma by GeneScreen ELISA for samples collected ≥18 months; or cell pellets by Amplicor HIV -1 DNA test version 1.5 (Roche Diagnostic Systems) for samples collected <18 months). If this sample was HIV-negative, the infant was classified as negative; if it was HIV-positive, samples collected at younger ages were tested to determine timing of infection.

Education and counseling about infant feeding in the context of HIV was updated throughout the trial. When the trial began, information about HIV transmission through breastfeeding was scanty. In June 1998, new infant feeding guidelines were published by UNAIDS/UNICEF/WHO stating that HIV-positive mothers should be fully informed about the risks and benefits of infant feeding alternatives and empowered to make their best personal choice. In response, we modified our procedures to provide 24-hour turn-around time for maternal HIV test results. Study nurses were trained to counsel HIV-positive women about feeding options and kitchens were established for teaching safe replacement feeding. Additional funding was obtained to conduct formative research to inform a more effective program to educate mothers about infant feeding in the context of HIV. This program included group education, incorporating infant feeding issues into individual counseling, and integrating mother to child HIV transmission issues into on-going work-site education programs targeting men, which were being run by other organizations in Harare. The program was fully implemented within the trial by November 1st 1999. It emphasized exclusive breastfeeding for HIV-positive mothers who chose to breastfeed, optimal breastfeeding techniques to avoid cracked nipples, milk stasis, and mastitis; prompt treatment of breast problems; and safe sex practices especially during the breastfeeding period. These four 'safer breastfeeding' practices were also promoted among all status-unknown and HIV negative women. Known HIV-positive women were counseled to stop breastfeeding early.

All laboratory analyses and data management was conducted in Harare. The protocol and interim analyses were reviewed by an external data safety and monitoring committee.

The study protocol was approved by the Medical Research Council of Zimbabwe, The Medicines Control Authority of Zimbabwe, The Johns Hopkins Bloomberg School of Public Health Committee on Human Research, and the Montreal General Hospital Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* mothers and their neonates delivering at a study recruitment site during the recruitment period

Exclusion Criteria:

* mother in intensive care unit
* mother not fully conscious
* maternal temperature > 39˚
* Mother is 'nil per mouth' (NPO)
* Mother is terminally ill as indicated in medical notes
* Infant is NPO
* Infant is terminally ill as indicated in medical notes
* Infant birth weight <1500 g
* Infant is a twin or triplet delivery
* Regular place of residence is outside Harare.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28220 (Actual)
Dates: Start 1997-11 (Actual); Primary Completion 2001-05 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
1. HIV infection rate among baseline HIV-negative babies born to HIV-positive mothers at 24 months | By 24 months of age
2. Infant mortality rate among all infants, infants born to HIV-negative mothers, and infants born to HIV-positive mothers at 6 months | by 12 months of age
3. HIV infection rates among baseline HIV-negative mothers at 24 months | by 24 months postpartum

SECONDARY OUTCOMES:
1. HIV infection or death rate among baseline HIV-negative babies born to HIV-positive mothers at 6, 12, and 18 months | By 24 months of age
2. HIV infection or death rate among 6-wk HIV-negative babies born to HIV-positive mothers at 6, 12, 18, 24 months | by 24 months of age
3. Serum and breast milk retinol concentration among women at 12 months | 12 months postpartum
4. Modified relative dose response ratios among infants at 6 wk, and 3, 6, 9, and 12 months. | 12 months post partum
5. Viral load among HIV-positive women at 6 wk, and 3, 6, 9, and 12 months. | 12 months postpartum
6. Weight for age among infants at 12 months | 12 months of age
7. Weight for length among infants at 12 months | 12 months of age
8. Length for age among infants at 12 months | 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Jean H Humphrey, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Pubic Health

REFERENCES:
- [Background] Humphrey JH, Rice AL. Vitamin A supplementation of young infants. Lancet. 2000 Jul 29;356(9227):422-4. doi: 10.1016/S0140-6736(00)02541-1. PMID 10972388
- [Background] Humphrey J, Iliff P. Is breast not best? Feeding babies born to HIV-positive mothers: bringing balance to a complex issue. Nutr Rev. 2001 Apr;59(4):119-27. doi: 10.1111/j.1753-4887.2001.tb06999.x. PMID 11368506
- [Background] Miller M, Humphrey J, Johnson E, Marinda E, Brookmeyer R, Katz J. Why do children become vitamin A deficient? J Nutr. 2002 Sep;132(9 Suppl):2867S-2880S. doi: 10.1093/jn/132.9.2867S. PMID 12221263
- [Background] Miller M, Iliff P, Stoltzfus RJ, Humphrey J. Breastmilk erythropoietin and mother-to-child HIV transmission through breastmilk. Lancet. 2002 Oct 19;360(9341):1246-8. doi: 10.1016/S0140-6736(02)11277-3. PMID 12401271
- [Background] Stoltzfus RJ, Humphrey JH. Vitamin A and the nursing mother-infant dyad: evidence for intervention. Adv Exp Med Biol. 2002;503:39-47. doi: 10.1007/978-1-4615-0559-4_4. PMID 12026026
- [Background] Humphrey JH, Quinn T, Fine D, Lederman H, Yamini-Roodsari S, Wu LS, Moeller S, Ruff AJ. Short-term effects of large-dose vitamin A supplementation on viral load and immune response in HIV-infected women. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Jan 1;20(1):44-51. doi: 10.1097/00042560-199901010-00007. PMID 9928729
- [Background] Iliff PJ, Humphrey JH, Mahomva AI, Zvandasara P, Bonduelle M, Malaba LC, Nathoo KJ. Tolerance of large doses of vitamin A given to mothers and their babies shortly after delivery. Nutr Res 1999; 19 (10): 1437-1446.
- [Background] Matte C, Lacaille J, Zijenah L, Ward B, Roger M. HLA-G and HLA-E polymorphisms in an indigenous African population. The ZVITAMBO Study Group. Hum Immunol. 2000 Nov;61(11):1150-6. doi: 10.1016/s0198-8859(00)00200-7. PMID 11137220
- [Background] Humphrey JH and Ichord RN: Safety of vitamin A supplementation of postpartum women and young children. Food and Nutrition Bulletin (2001) 22: 311-319.
- [Background] Matte C, Lacaille J, Zijenah L, Ward B, Roger M; ZVITAMBO Study Group. HLA-G exhibits low level of polymorphism in indigenous East Africans. Hum Immunol. 2002 Jun;63(6):495-501. doi: 10.1016/s0198-8859(02)00391-9. PMID 12039526
- [Background] Lajoie J, Zijenah LS, Faucher MC, Ward BJ, Roger M; ZVITAMBO Study Group. New transporter associated with antigen processing (TAP-2) polymorphisms in the Shona people of Zimbabwe. Hum Immunol. 2003 Jul;64(7):733-40. doi: 10.1016/s0198-8859(03)00079-x. PMID 12826376
- [Background] Lajoie J, Zijenah LS, Faucher MC, Ward BJ, Roger M; ZVITAMBO Study Group. Novel TAP1 polymorphisms in indigenous Zimbabweans: their potential implications on TAP function and in human diseases. Hum Immunol. 2003 Aug;64(8):823-9. doi: 10.1016/s0198-8859(03)00110-1. PMID 12878362
- [Background] Rollins N, Meda N, Becquet R, Coutsoudis A, Humphrey J, Jeffrey B, Kanshana S, Kuhn L, Leroy V, Mbori-Ngacha D, McIntyre J, Newell ML; Ghent IAS Working Group on HIV in Women and Children. Preventing postnatal transmission of HIV-1 through breast-feeding: modifying infant feeding practices. J Acquir Immune Defic Syndr. 2004 Feb 1;35(2):188-95. doi: 10.1097/00126334-200402010-00014. PMID 14722453
- [Background] Lajoie J, Hargrove J, Zijenah LS, Humphrey JH, Ward BJ, Roger M. Genetic variants in nonclassical major histocompatibility complex class I human leukocyte antigen (HLA)-E and HLA-G molecules are associated with susceptibility to heterosexual acquisition of HIV-1. J Infect Dis. 2006 Jan 15;193(2):298-301. doi: 10.1086/498877. Epub 2005 Dec 1. PMID 16362895
- [Background] Miller MF, Humphrey JH, Iliff PJ, Malaba LC, Mbuya NV, Stoltzfus RJ; ZVITAMBO Study Group. Neonatal erythropoiesis and subsequent anemia in HIV-positive and HIV-negative Zimbabwean babies during the first year of life: a longitudinal study. BMC Infect Dis. 2006 Jan 3;6:1. doi: 10.1186/1471-2334-6-1. PMID 16390553
- [Background] Humphrey JH, Iliff PJ, Marinda E, Mutasa K, Moulton LH, Chidawanyika H, Ward BJ, Nathoo KJ, Malaba LC, Zijenah LS, Zvandasara P, Ntozini R, Mzengeza F, Mahomva A, Ruff A, Mbizvo M, Zunguza C, and the ZVITAMBO Study Group: Impact of single large doses of vitamin A given during the postpartum period to HIV-infected women and their neonates on breastfeeding-associated mother-to-child-transmission of HIV and infant mortality in Zimbabwe. J Infectious Diseases 2006, 193:860-871. Selected for an editorial: Fawzi, WW: The benefits and concerns related to vitamin A supplementation. J Infectious Diseases 2006;193:756-9.
- [Background] Humphrey JH, Hargrove JW, Malaba LC, Iliff PJ, Moulton LH, Mutasa K, Zvandasara P, Nathoo KJ, Mzengeza F, Chidawanyika H, Zijenah LS, Ward BJ; ZVITAMBO Study Group. HIV incidence among post-partum women in Zimbabwe: risk factors and the effect of vitamin A supplementation. AIDS. 2006 Jun 26;20(10):1437-46. doi: 10.1097/01.aids.0000233578.72091.09. PMID 16791019
- [Background] Zvandasara P, Hargrove JW, Ntozini R, Chidawanyika H, Mutasa K, Iliff PJ, Moulton LH, Mzengeza F, Malaba LC, Ward BJ, Nathoo KJ, Zijenah LS, Mbizvo M, Zunguza C, Humphrey JH; ZVITAMBO Study Group. Mortality and morbidity among postpartum HIV-positive and HIV-negative women in Zimbabwe: risk factors, causes, and impact of single-dose postpartum vitamin A supplementation. J Acquir Immune Defic Syndr. 2006 Sep;43(1):107-16. doi: 10.1097/01.qai.0000229015.77569.c7. PMID 16885772
- [Background] Miller MF, Stoltzfus RJ, Iliff PJ, Malaba LC, Mbuya NV; Zimbabwe Vitamin A for Mothers and Babies Project (ZVITAMBO) Study Group; Humphrey JH. Effect of maternal and neonatal vitamin A supplementation and other postnatal factors on anemia in Zimbabwean infants: a prospective, randomized study. Am J Clin Nutr. 2006 Jul;84(1):212-22. doi: 10.1093/ajcn/84.1.212. PMID 16825698
- [Background] Piwoz EG, Humphrey JH, Tavengwa NV, Iliff PJ, Marinda ET, Zunguza CD, Nathoo KJ, Mutasa K, Moulton LH, Ward BJ. The impact of safer breastfeeding practices on postnatal HIV-1 transmission in Zimbabwe. Am J Public Health. 2007 Jul;97(7):1249-54. doi: 10.2105/AJPH.2006.085704. Epub 2007 May 30. PMID 17538064
- [Background] Tavengwa NV, Piwoz EG, Iliff PJ, Moulton LH, Zunguza CD, Nathoo KJ, Hargrove JW; ZVITAMBO Study Group; Humphrey JH. Adoption of safer infant feeding and postpartum sexual practices and their relationship to maternal HIV status and risk of acquiring HIV in Zimbabwe. Trop Med Int Health. 2007 Jan;12(1):97-106. doi: 10.1111/j.1365-3156.2006.01758.x. PMID 17207153
- [Background] Piwoz EG, Humphrey JH, Marinda ET, Mutasa K, Moulton LH, Iliff PJ. Effects of infant sex on mother-to-child transmission of HIV-1 according to timing of infection in Zimbabwe. AIDS. 2006 Oct 3;20(15):1981-4. doi: 10.1097/01.aids.0000247123.04703.6e. PMID 16988523
- [Background] Marinda E, Humphrey JH, Iliff PJ, Mutasa K, Nathoo KJ, Piwoz EG, Moulton LH, Salama P, Ward BJ; ZVITAMBO Study Group. Child mortality according to maternal and infant HIV status in Zimbabwe. Pediatr Infect Dis J. 2007 Jun;26(6):519-26. doi: 10.1097/01.inf.0000264527.69954.4c. PMID 17529870
- [Background] Humphrey JH, Nathoo KJ, Hargrove JW, Iliff PJ, Mutasa KE, Moulton LH, Chidawanyika H, Malaba LC, Zijenah LS, Zvandasara P, Ntozini R, Zunguza CD, Ward BJ; ZVITAMBO Study Group. HIV-1 and HIV-2 prevalence and associated risk factors among postnatal women in Harare, Zimbabwe. Epidemiol Infect. 2007 Aug;135(6):933-42. doi: 10.1017/S0950268806007709. Epub 2007 Jan 12. PMID 17217549
- [Background] Hargrove JW, Humphrey JH, Mutasa K, Parekh BS, McDougal JS, Ntozini R, Chidawanyika H, Moulton LH, Ward B, Nathoo K, Iliff PJ, Kopp E. Improved HIV-1 incidence estimates using the BED capture enzyme immunoassay. AIDS. 2008 Feb 19;22(4):511-8. doi: 10.1097/QAD.0b013e3282f2a960. PMID 18301064
- [Background] Cowan FM, Humphrey JH, Ntozini R, Mutasa K, Morrow R, Iliff P. Maternal Herpes simplex virus type 2 infection, syphilis and risk of intra-partum transmission of HIV-1: results of a case control study. AIDS. 2008 Jan 11;22(2):193-201. doi: 10.1097/QAD.0b013e3282f2a939. PMID 18097221
- [Background] Lunney KM, Jenkins AL, Tavengwa NV, Majo F, Chidhanguro D, Iliff P, Strickland GT, Piwoz E, Iannotti L, Humphrey JH. HIV-positive poor women may stop breast-feeding early to protect their infants from HIV infection although available replacement diets are grossly inadequate. J Nutr. 2008 Feb;138(2):351-7. doi: 10.1093/jn/138.2.351. PMID 18203903
- [Background] Rawat R, Stoltzfus RJ, Ntozini R, Mutasa K, Iliff PJ, Humphrey JH. Influence of inflammation as measured by alpha-1-acid glycoprotein on iron status indicators among HIV-positive postpartum Zimbabwean women. Eur J Clin Nutr. 2009 Jun;63(6):787-93. doi: 10.1038/ejcn.2008.33. Epub 2008 May 28. PMID 18506200
- [Background] Iliff P, Ntozini R, Nathoo K, Piwoz E, Moulton L; ZVITAMBO Study Group; Humphrey J. Making a working clinical diagnosis of HIV infection in infants in Zimbabwe. Trop Med Int Health. 2008 Dec;13(12):1459-69. doi: 10.1111/j.1365-3156.2008.02178.x. PMID 19055624
- [Background] Rawat R, Humphrey JH, Ntozini R, Mutasa K, Iliff PJ, Stoltzfus RJ. Elevated iron stores are associated with HIV disease severity and mortality among postpartum women in Zimbabwe. Public Health Nutr. 2009 Sep;12(9):1321-9. doi: 10.1017/S136898000800390X. Epub 2008 Nov 12. PMID 19000344
- [Background] Koyanagi A, Humphrey JH, Moulton LH, Ntozini R, Mutasa K, Iliff P, Black RE. Effect of early exclusive breastfeeding on morbidity among infants born to HIV-negative mothers in Zimbabwe. Am J Clin Nutr. 2009 May;89(5):1375-82. doi: 10.3945/ajcn.2008.26810. Epub 2009 Apr 1. PMID 19339398
- [Background] Boily-Larouche G, Iscache AL, Zijenah LS, Humphrey JH, Mouland AJ, Ward BJ, Roger M. Functional genetic variants in DC-SIGNR are associated with mother-to-child transmission of HIV-1. PLoS One. 2009 Oct 7;4(10):e7211. doi: 10.1371/journal.pone.0007211. PMID 19809496
- [Background] Lunney KM, Iliff P, Mutasa K, Ntozini R, Magder LS, Moulton LH, Humphrey JH. Associations between breast milk viral load, mastitis, exclusive breast-feeding, and postnatal transmission of HIV. Clin Infect Dis. 2010 Mar 1;50(5):762-9. doi: 10.1086/650535. PMID 20121424
- [Background] Koyanagi A, Ruff AJ, Moulton LH, Ntozini R, Mutasa K, Iliff P, Humphrey JH; ZVITAMBO Study Group. Postpartum plasma CD4 change in HIV-positive women: implications for timing of HAART initiation. AIDS Res Hum Retroviruses. 2010 May;26(5):547-52. doi: 10.1089/aid.2009.0138. PMID 20455759
- [Background] Hargrove JW, Humphrey JH; ZVITAMBO Study Group. Mortality among HIV-positive postpartum women with high CD4 cell counts in Zimbabwe. AIDS. 2010 Jan 28;24(3):F11-4. doi: 10.1097/qad.0b013e328335749d. PMID 20095074
- [Background] Hargrove J, Humphrey J; ZVITAMBO Study Group. Short communication: Simplified estimation of the long-term specificity of the BED assay to improve estimates of HIV incidence. AIDS Res Hum Retroviruses. 2010 Sep;26(9):977-9. doi: 10.1089/aid.2010.0009. PMID 20718627
- [Background] Williams BG, Hargrove JW, Humphrey JH. The benefits of early treatment for HIV. AIDS. 2010 Jul 17;24(11):1790-1. doi: 10.1097/QAD.0b013e32833ac860. No abstract available. PMID 20588108
- [Background] Rawat R, Humphrey JH, Mutasa K, Ntozini R, Stoltzfus RJ. Short communication: predicting adverse HIV-related outcomes in a resource-limited setting: use of the inflammation marker alpha(1)-acid glycoprotein. AIDS Res Hum Retroviruses. 2010 Nov;26(11):1171-4. doi: 10.1089/aid.2010.0053. Epub 2010 Oct 26. PMID 20977355
- [Background] Koyanagi A, Humphrey JH, Ntozini R, Nathoo K, Moulton LH, Iliff P, Mutasa K, Ruff A, Ward B; ZVITAMBO Study Group. Morbidity among human immunodeficiency virus-exposed but uninfected, human immunodeficiency virus-infected, and human immunodeficiency virus-unexposed infants in Zimbabwe before availability of highly active antiretroviral therapy. Pediatr Infect Dis J. 2011 Jan;30(1):45-51. doi: 10.1097/INF.0b013e3181ecbf7e. PMID 21173675
- [Background] Humphrey JH, Marinda E, Mutasa K, Moulton LH, Iliff PJ, Ntozini R, Chidawanyika H, Nathoo KJ, Tavengwa N, Jenkins A, Piwoz EG, Van de Perre P, Ward BJ; ZVITAMBO study group. Mother to child transmission of HIV among Zimbabwean women who seroconverted postnatally: prospective cohort study. BMJ. 2010 Dec 22;341:c6580. doi: 10.1136/bmj.c6580. PMID 21177735
- [Background] Kirkwood B, Humphrey J, Moulton L, Martines J. Neonatal vitamin A supplementation and infant survival. Lancet. 2010 Nov 13;376(9753):1643-4. doi: 10.1016/S0140-6736(10)61895-8. Epub 2010 Oct 13. No abstract available. PMID 20950849
- [Background] Hargrove JW, Humphrey JH, Mahomva A, Williams BG, Chidawanyika H, Mutasa K, Marinda E, Mbizvo MT, Nathoo KJ, Iliff PJ, Mugurungi O; ZVITAMBO Study Group. Declining HIV prevalence and incidence in perinatal women in Harare, Zimbabwe. Epidemics. 2011 Jun;3(2):88-94. doi: 10.1016/j.epidem.2011.02.004. Epub 2011 Mar 2. PMID 21624779
- [Background] Koyanagi A, Humphrey JH, Moulton LH, Ntozini R, Mutasa K, Iliff P, Ruff AJ; Zvitambo Study Group. Predictive value of weight loss on mortality of HIV-positive mothers in a prolonged breastfeeding setting. AIDS Res Hum Retroviruses. 2011 Nov;27(11):1141-8. doi: 10.1089/AID.2010.0293. Epub 2011 Feb 16. PMID 21226627
- [Background] Marinda ET, Moulton LH, Humphrey JH, Hargrove JW, Ntozini R, Mutasa K, Levin J. In utero and intra-partum HIV-1 transmission and acute HIV-1 infection during pregnancy: using the BED capture enzyme-immunoassay as a surrogate marker for acute infection. Int J Epidemiol. 2011 Aug;40(4):945-54. doi: 10.1093/ije/dyr055. Epub 2011 Apr 5. PMID 21471020
- [Background] Mutasa K, Ntozini R, Prendergast A, Iliff P, Rukobo S, Moulton LH, Ward BJ, Humphrey JH; ZVITAMBO Study Group. Impact of six-week viral load on mortality in HIV-infected Zimbabwean infants. Pediatr Infect Dis J. 2012 Sep;31(9):948-50. doi: 10.1097/INF.0b013e318266aac2. PMID 22743826
- [Background] Gumbo H, Chasekwa B, Church JA, Ntozini R, Mutasa K, Humphrey JH, Prendergast AJ. Congenital and postnatal CMV and EBV acquisition in HIV-infected Zimbabwean infants. PLoS One. 2014 Dec 18;9(12):e114870. doi: 10.1371/journal.pone.0114870. eCollection 2014. PMID 25522217
- [Background] Mupfudze TG, Stoltzfus RJ, Rukobo S, Moulton LH, Humphrey JH, Prendergast AJ; SHINE Trial Team; Jones AD, Manges A, Mangwadu G, Maluccio JA, Mbuya MN, Ntozini R, Tielsch JM. Plasma Concentrations of Hepcidin in Anemic Zimbabwean Infants. PLoS One. 2015 Aug 7;10(8):e0135227. doi: 10.1371/journal.pone.0135227. eCollection 2015. PMID 26252205
- [Background] Evans C, Chasekwa B, Ntozini R, Humphrey JH, Prendergast AJ. Head circumferences of children born to HIV-infected and HIV-uninfected mothers in Zimbabwe during the preantiretroviral therapy era. AIDS. 2016 Sep 24;30(15):2323-8. doi: 10.1097/QAD.0000000000001196. PMID 27428746
- [Background] Gough EK, Moodie EE, Prendergast AJ, Ntozini R, Moulton LH, Humphrey JH, Manges AR. Linear growth trajectories in Zimbabwean infants. Am J Clin Nutr. 2016 Dec;104(6):1616-1627. doi: 10.3945/ajcn.116.133538. Epub 2016 Nov 2. PMID 27806980
- [Background] Evans C, Chasekwa B, Rukobo S, Govha M, Mutasa K, Ntozini R, Humphrey JH, Prendergast AJ. Cytomegalovirus Acquisition and Inflammation in Human Immunodeficiency Virus-Exposed Uninfected Zimbabwean Infants. J Infect Dis. 2017 Mar 1;215(5):698-702. doi: 10.1093/infdis/jiw630. PMID 28011912
- [Background] Omoni AO, Ntozini R, Evans C, Prendergast AJ, Moulton LH, Christian PS, Humphrey JH. Child Growth According to Maternal and Child HIV Status in Zimbabwe. Pediatr Infect Dis J. 2017 Sep;36(9):869-876. doi: 10.1097/INF.0000000000001574. PMID 28198792
- [Result] Zijenah LS, Humphrey J, Nathoo K, Malaba L, Zvandasara P, Mahomva A, Iliff P, Mbizvo MT. Evaluation of the prototype Roche DNA amplification kit incorporating the new SSK145 and SKCC1B primers in detection of human immunodeficiency virus type 1 DNA in Zimbabwe. J Clin Microbiol. 1999 Nov;37(11):3569-71. doi: 10.1128/JCM.37.11.3569-3571.1999. PMID 10523553
- [Result] Zijenah LS, Moulton LH, Iliff P, Nathoo K, Munjoma MW, Mutasa K, Malaba L, Zvandasara P, Ward BJ, Humphrey J; ZVITAMBO Study Group. Timing of mother-to-child transmission of HIV-1 and infant mortality in the first 6 months of life in Harare, Zimbabwe. AIDS. 2004 Jan 23;18(2):273-80. doi: 10.1097/00002030-200401230-00017. PMID 15075545
- [Result] Malaba LC, Iliff PJ, Nathoo KJ, Marinda E, Moulton LH, Zijenah LS, Zvandasara P, Ward BJ, Humphrey JH; ZVITAMBO Study Group. Effect of postpartum maternal or neonatal vitamin A supplementation on infant mortality among infants born to HIV-negative mothers in Zimbabwe. Am J Clin Nutr. 2005 Feb;81(2):454-60. doi: 10.1093/ajcn.81.2.454. PMID 15699235
- [Result] Iliff PJ, Piwoz EG, Tavengwa NV, Zunguza CD, Marinda ET, Nathoo KJ, Moulton LH, Ward BJ, Humphrey JH; ZVITAMBO study group. Early exclusive breastfeeding reduces the risk of postnatal HIV-1 transmission and increases HIV-free survival. AIDS. 2005 Apr 29;19(7):699-708. doi: 10.1097/01.aids.0000166093.16446.c9. PMID 15821396
- [Result] Piwoz EG, Iliff PJ, Tavengwa N, Gavin L, Marinda E, Lunney K, Zunguza C, Nathoo KJ, Humphrey JH. An education and counseling program for preventing breast-feeding-associated HIV transmission in Zimbabwe: design and impact on maternal knowledge and behavior. J Nutr. 2005 Apr;135(4):950-5. doi: 10.1093/jn/135.4.950. PMID 15795468
- [Result] Miller MF, Stoltzfus RJ, Mbuya NV, Malaba LC, Iliff PJ, Humphrey JH; ZVITAMBO Study Group. Total body iron in HIV-positive and HIV-negative Zimbabwean newborns strongly predicts anemia throughout infancy and is predicted by maternal hemoglobin concentration. J Nutr. 2003 Nov;133(11):3461-8. doi: 10.1093/jn/133.11.3461. PMID 14608059
- [Derived] Church JA, Rukobo S, Govha M, Carmolli MP, Diehl SA, Chasekwa B, Ntozini R, Mutasa K, Humphrey JH, Kirkpatrick BD, Prendergast AJ. Neonatal vitamin A supplementation and immune responses to oral polio vaccine in Zimbabwean infants. Trans R Soc Trop Med Hyg. 2019 Mar 1;113(3):110-115. doi: 10.1093/trstmh/try126. PMID 30576507